CLINICAL TRIAL: NCT06066307
Title: Olfactory Performance in Culinary Arts Students
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leigh Sowerby (Other)
Collaborators: Fanshawe College (Unknown)
Responsible Party: Sponsor-Investigator, Leigh Sowerby, MD, MHM, FRCSC, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 23-06-11-1
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Loss of Smell; Olfactory Disorder
Keywords: Olfactory training; Olfaction; Smell; Hyposmia; Anosmia; Olfactory Disfunction
MeSH Terms: conditions — Anosmia | interventions — Olfactory Training

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Research staff involved in the smell tests and questionnaires administration will not be aware of the subjects allocation (whether OT or control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Olfactory training - Culinary arts students (Experimental): Students in culinary skill training program will perform olfactory training by sniffing four specific essential oils twice daily, over the entire semester (4-month period). The odors will comprise four major odor categories: flowery (phenyl ethyl alcohol/rose), aromatic (eucalyptol), fruity (citronellal/lemon), and resinous (eugenol). They will be assessed before and after the school semester.
  Interventions: Other: Olfactory training
- Control group - Culinary arts students (No Intervention): Students in culinary skill training program will be assessed before and after the school semester, without any intervention throughout this period.
- Olfactory training - Information Technology students (Experimental): Students in Information Technology program will perform olfactory training by sniffing four specific essential oils twice daily, over the entire semester (4-month period). The odors will comprise four major odor categories: flowery (phenyl ethyl alcohol/rose), aromatic (eucalyptol), fruity (citronellal/lemon), and resinous (eugenol). They will be assessed before and after the school semester.
  Interventions: Other: Olfactory training
- Control group - Information Technology students (No Intervention): Students in Information Technology program will be assessed before and after the school semester, without any intervention throughout this period.

INTERVENTIONS:
Other: Olfactory training — Olfactory training will be performed by sniffing four specific essential oils twice daily for 30 seconds each. Participants are encouraged to visualize the item they are smelling, while they perform the procedure, in a quiet room, with their eyes closed. The odors will comprise four major odor categories: flowery (phenyl ethyl alcohol/rose), aromatic (eucalyptol), fruity (citronellal/lemon), and resinous (eugenol).
  Other Names: Smell training; Smell Rehabilitation; Olfactory Rehabilitation
  Arms: Olfactory training - Culinary arts students; Olfactory training - Information Technology students

SUMMARY:
The COVID-19 pandemic brought impaired smell and taste to the forefront of international public awareness and clinical importance. Loss of smell can impair awareness of environmental hazards, alter appetite, and have negative effects on social behavior and well-being. Despite the significant functional impact associated with impaired olfaction, few effective treatments are available. Olfactory training (OT), the mainstay of treatment, is a self-administered therapy which involves a routine of repetitive brief odor exposures over several weeks. The process has been shown to improve odor discrimination, identification and detection threshold. However, the structured design and daily time commitment may be difficult to adopt for some patients, leading to poor compliance. Moreover, OT only exposes patients to a limited number of odours, failing to replicate the complexity of odor mixtures experienced daily in our chemosensory environment. OT has mainly been studied with four conventional odours encompassing the major odor categories; phenyl ethyl alcohol/rose (flowery odor), eucalyptol (aromatic), citronellal/lemon (fruity), and eugenol (clove) (resinous); however, this neglects the importance of emphasizing odors that culturally specific or personally relevant to the patient. For some patients, these factors could hinder their ability to adopt and comply with therapy.

In contrast, cooking is a culturally ubiquitous activity that is already performed daily by most people, and naturally exposes us to personally meaningful and culturally relevant odors. However, there have been no published studies investigating the impact that odors encountered during meal preparation have on olfactory performance and development. The present study aims to compare the olfactory effects of culinary skills training to those of a conventionally designed OT program. To achieve this, olfactory testing will be conducted on students enrolled in a professional culinary skills training program at Fanshawe College, and a control group consisting of students in non-olfactory dependent programs at the same institution. To compare the effect of cooking to conventional OT, the study will be repeated for a second semester and students will be asked to perform concurrent OT.

DETAILED DESCRIPTION:
This factorially designed randomized control trial is designed to compare the effects of a culinary skills training program to a typical olfactory training program on olfactory ability, awareness, and quality of life. Students enrolled in a culinary skills training program and those in a different discipline with no relevant dependence on olfactory function (information technology) will have their olfactory performance assessed before and after the completion of the program semester. The investigators will then repeat the experiment in the subsequent semester with a new group of students, asking them to perform routine OT throughout the semester.

Objective olfactory assessment will be performed with the Sniffin'Sticks olfactory test kit (Burghart, Wedel, Germany). Additionally, they will be asked to complete questionnaires that evaluate their olfactory awareness, the 32-item Odor Awareness Scale. The study aims to compare the effect of routine exposure to the chemosensory environment of cooking with conventional odor training (OT) in improving olfactory function.

Hypothesis and Objectives Objective 1: To compare the effect of culinary skill training to a control group on objective olfactory performance, subjective olfactory awareness and olfactory related quality of life.

* Hypothesis 1: Participants who complete a semester of culinary skill training will experience improvements in odor threshold discrimination identification scores compared to students studying in non-chemosensory dependent fields.
* Hypothesis 2: Participants who complete a semester of culinary skill training will experience improvements in subjective odor awareness compared to students studying in non- chemosensory dependent fields.
* Hypothesis 3: Participants who complete a semester of culinary skill training will experience improvements in olfactory specific quality of life compared to students studying in non- chemosensory dependent fields.

Objective 2: To compare the effect of culinary skill training with OT to conventional OT on objective olfactory performance, subjective olfactory awareness and olfactory related quality of life

* Hypothesis 1: Participants who complete a semester of culinary skill training with OT will experience further improvements in odor their threshold discrimination identification scores.
* Hypothesis 2: Participants who complete a semester of culinary skill training with OT will experience improvements in subjective odor awareness that are greater in magnitude to the improvements gained by participants practicing OT.
* Hypothesis 3: Participants who complete a semester of culinary skill training with OT will experience improvements in olfactory specific quality of life that are greater in magnitude to the improvements gained by participants practicing OT.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* enrolled in an introductory training program at Fanshawe collage (Culinary arts or Information Technology)
* capable of providing informed written consent
* capable of reading and writing in English

Exclusion Criteria:

* Participants with a history of anosmia, and chronic sinus disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-11-21 (Estimated)

PRIMARY OUTCOMES:
Odor threshold discrimination identification scores | Baseline, 4 months (after school semester)
  Changes from Baseline (before the school semester) on Sniffin Stick test scores considering the three olfactory dimensions (threshold, discrimination, and identification). Higher scores in this test mean better olfactory status.

SECONDARY OUTCOMES:
Subjective odor awareness | Baseline, 4 months (after school semester)
  Changes from Baseline (before the school semester) on the Odor Awareness Scale. The Odor Awareness Scale questionnaire evaluates the effects of odors on attention, emotion, memory, product purchase, and the sensitivity and importance of odors. This questionnaire broadly covers odor situations pertaining to eating, drinking, nature, and social interactions. Higher scores in this test mean better olfactory status and better odor awareness.
Olfactory specific quality of life | Baseline, 4 months (after school semester)
  Changes from Baseline (before the school semester) on the Odor Awareness Scale. The Odor Awareness Scale questionnaire evaluates the effects of odors on attention, emotion, memory, product purchase, and the sensitivity and importance of odors. This questionnaire broadly covers odor situations pertaining to eating, drinking, nature, and social interactions. Higher scores in this test mean better olfactory status and better olfactory-specific quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Fanshawe College, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yan CH, Faraji F, Prajapati DP, Boone CE, DeConde AS. Association of chemosensory dysfunction and COVID-19 in patients presenting with influenza-like symptoms. Int Forum Allergy Rhinol. 2020 Jul;10(7):806-813. doi: 10.1002/alr.22579. Epub 2020 Jun 1. PMID 32279441
- [Background] Pence TS, Reiter ER, DiNardo LJ, Costanzo RM. Risk factors for hazardous events in olfactory-impaired patients. JAMA Otolaryngol Head Neck Surg. 2014 Oct;140(10):951-5. doi: 10.1001/jamaoto.2014.1675. PMID 25170573
- [Background] McCrickerd K, Forde CG. Sensory influences on food intake control: moving beyond palatability. Obes Rev. 2016 Jan;17(1):18-29. doi: 10.1111/obr.12340. Epub 2015 Dec 11. PMID 26662879
- [Background] Boesveldt S, Parma V. The importance of the olfactory system in human well-being, through nutrition and social behavior. Cell Tissue Res. 2021 Jan;383(1):559-567. doi: 10.1007/s00441-020-03367-7. Epub 2021 Jan 12. PMID 33433688
- [Background] Philpott CM, Boak D. The impact of olfactory disorders in the United kingdom. Chem Senses. 2014 Oct;39(8):711-8. doi: 10.1093/chemse/bju043. Epub 2014 Sep 8. PMID 25201900
- [Background] Hummel T, Rissom K, Reden J, Hahner A, Weidenbecher M, Huttenbrink KB. Effects of olfactory training in patients with olfactory loss. Laryngoscope. 2009 Mar;119(3):496-9. doi: 10.1002/lary.20101. PMID 19235739
- [Background] Pekala K, Chandra RK, Turner JH. Efficacy of olfactory training in patients with olfactory loss: a systematic review and meta-analysis. Int Forum Allergy Rhinol. 2016 Mar;6(3):299-307. doi: 10.1002/alr.21669. Epub 2015 Dec 1. PMID 26624966
- [Background] Hummel T, Whitcroft KL, Andrews P, Altundag A, Cinghi C, Costanzo RM, Damm M, Frasnelli J, Gudziol H, Gupta N, Haehne A, Holbrook E, Hong SC, Hornung D, Huttenbrink KB, Kamel R, Kobayashi M, Konstantinidis I, Landis BN, Leopold DA, Macchi A, Miwa T, Moesges R, Mullol J, Mueller CA, Ottaviano G, Passali GC, Philpott C, Pinto JM, Ramakrishnan VJ, Rombaux P, Roth Y, Schlosser RA, Shu B, Soler G, Stjarne P, Stuck BA, Vodicka J, Welge-Luessen A. Position paper on olfactory dysfunction. Rhinol Suppl. 2017 Mar;54(26):1-30. doi: 10.4193/Rhino16.248. PMID 29528615
- [Background] Fornazieri MA, Garcia ECD, Lopes NMD, Miyazawa INI, Silva GDS, Monteiro RDS, Pinna FR, Voegels RL, Doty RL. Adherence and Efficacy of Olfactory Training as a Treatment for Persistent Olfactory Loss. Am J Rhinol Allergy. 2020 Mar;34(2):238-248. doi: 10.1177/1945892419887895. Epub 2019 Nov 25. No abstract available. PMID 31766853
- [Background] Altundag A, Cayonu M, Kayabasoglu G, Salihoglu M, Tekeli H, Saglam O, Hummel T. Modified olfactory training in patients with postinfectious olfactory loss. Laryngoscope. 2015 Aug;125(8):1763-6. doi: 10.1002/lary.25245. Epub 2015 Jun 2. PMID 26031472
- [Background] Greenberg MI, Curtis JA, Vearrier D. The perception of odor is not a surrogate marker for chemical exposure: a review of factors influencing human odor perception. Clin Toxicol (Phila). 2013 Feb;51(2):70-6. doi: 10.3109/15563650.2013.767908. PMID 23387344
- [Background] Majid A. Human Olfaction at the Intersection of Language, Culture, and Biology. Trends Cogn Sci. 2021 Feb;25(2):111-123. doi: 10.1016/j.tics.2020.11.005. Epub 2020 Dec 18. PMID 33349546
- [Background] Huisman JLA, Majid A. Psycholinguistic variables matter in odor naming. Mem Cognit. 2018 May;46(4):577-588. doi: 10.3758/s13421-017-0785-1. PMID 29435824
- [Background] Spence C. Perceptual learning in the chemical senses: A review. Food Res Int. 2019 Sep;123:746-761. doi: 10.1016/j.foodres.2019.06.005. Epub 2019 Jun 5. PMID 31285024